CLINICAL TRIAL: NCT02736474
Title: Effect of Naltrexone and Bupropion Combination on Weight Loss and Smoking Cessation in Obese, Cigarette-smoking Patients With Schizophrenia
Brief Title: Naltrexone and Bupropion Combination on Obese,Smoking Patients With Schizophrenia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Collaborators: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, DU, Jiang, Chief Physician, Shanghai Mental Health Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MZhao-005
Record Dates: First submitted 2016-03-23; First posted 2016-04-13 (Estimated); Results first posted 2021-10-22 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-09

CONDITIONS: Obese; Cigarette-smoking; Schizophrenia
MeSH Terms: conditions — Obesity; Cigarette Smoking; Schizophrenia | interventions — Naltrexone; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Naltrexone and Bupropion (Experimental): Naltrexone 3 tablets（15mg） once per day and Bupropion 1 capsule（150mg） once per day in the first two weeks. Then Naltrexone 5 tablets（25mg） once per day and Bupropion 2 capsules（300mg） once per day during the rest of the study.
  Interventions: Drug: Naltrexone; Drug: Bupropion
- Placebo Naltrexone and Bupropion (Placebo Comparator): Placebo Naltrexone 3 tablets+Placebo Bupropion 1 capsule once per day in the first two weeks. Then Placebo Naltrexone 5 tablets+Placebo Bupropion 2 capsule once per day during the rest of the study.
  Interventions: Drug: Placebo Naltrexone; Drug: Placebo Bupropion

INTERVENTIONS:
Drug: Naltrexone — 3 tablets（15mg） once per day in the first two weeks，then Naltrexone 5 tablets（25mg） once per day during the rest of the study.
  Arms: Naltrexone and Bupropion
Drug: Placebo Naltrexone — Placebo Naltrexone created and masked by the pharmacy to be used as a control.
  Arms: Placebo Naltrexone and Bupropion
Drug: Bupropion — 1 capsule（150mg） once per day in the first two weeks，then 2 capsules（300mg） once per day during the rest of the study.
  Arms: Naltrexone and Bupropion
Drug: Placebo Bupropion — Placebo Bupropion created and masked by the pharmacy to be used as a control.
  Arms: Placebo Naltrexone and Bupropion

SUMMARY:
The purpose of this research is to observe the efficacy of Naltrexone and Bupropion combination on weight loss and smoking cessation from baseline to week 24 compare to placebo.

DETAILED DESCRIPTION:
This is a randomized, double-blind, and placebo-controlled study. Subjects with evaluation and confirmation that inclusion and exclusion criteria are met, will be treated with naltrexone sustained release 15mg once per day and bupropion sustained release 150mg once per day in the first two weeks, and naltrexone 25mg once per day and bupropion 300mg once per day during the rest of the study.The purpose of this research is to observe the efficacy of Naltrexone and Bupropion on weight loss and smoking cessation compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia by the International Classification of Diseases 10th Revision (ICD-10);
* age between 18 and 65 years old;
* on stable antipsychotic medication treatment for at least one month;
* BMI > 28 kg/m2 according to BMI criterion for obesity in the Chinese population ， or BMI>27 kg/m2 in the presence of dyslipidemia, or male with waist circumference over 90cm;
* smoking at least 10 cigarettes daily for one year or longer;
* desire to lose weight and quit smoking.

Exclusion Criteria:

* Binge eating or other eating disorders;
* Current use of weight loss or antidiabetic medications;
* Current substance use (except nicotine or caffeine);
* Elevated hepatic transaminase levels (>2.5x normal range);
* Clinically significant Thyroid Stimulating Hormone（TSH） and/or thyroxine4（T4） abnormalities;
* History of seizure disorder;
* History of unstable cardiac problems or other unstable medication conditions;
* Being pregnant or nursing (for women).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Du, PhD, Principal Investigator — Chief Physician

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lyu X, Du J, Zhan G, Wu Y, Su H, Zhu Y, Jarskog F, Zhao M, Fan X. Naltrexone and Bupropion Combination Treatment for Smoking Cessation and Weight Loss in Patients With Schizophrenia. Front Pharmacol. 2018 Mar 5;9:181. doi: 10.3389/fphar.2018.00181. eCollection 2018. PMID 29563871

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Started | 11 | 11
Completed | 11 | 10
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.3 (5.7) | 54.1 (8.4) | 54.2 (7.0)
Sex/Gender, Customized [Number; unit: participants]
  male | 11 | 11 | 22
Race/Ethnicity, Customized [Number; unit: participants]
  Han | 11 | 11 | 22
Region of Enrollment [Number; unit: participants]
  China | 11 | 11 | 22
illness time duration [Mean (Standard Deviation); unit: years] | 29.8 (4.6) | 25.9 (9.1) | 27.9 (7.8)
smoking time duration [Mean (Standard Deviation); unit: years] | 28.6 (7.9) | 29.8 (9.8) | 29.2 (8.7)
breath CO level [Mean (Standard Deviation); unit: ppm] | 27.1 (23.2) | 27.7 (15.6) | 27.4 (19.3)
number of cigarettes smoked per week [Mean (Standard Deviation); unit: cigarettes per week] | 72.5 (5.7) | 77.6 (21.1) | 75.1 (15.3)
smoking craving [Mean (Standard Deviation); unit: units on a scale] — The visual analogue scale is a scale that is used to gauge smoking craving. Patients can choose a number from 0 to 10 to show their smoking craving, in which "0" represents "no craving" and "10" represents "intense urge".
  units on a scale | 6.3 (1.0) | 7.0 (1.4) | 6.6 (1.3)
body weight [Mean (Standard Deviation); unit: kg] | 74.7 (11.8) | 80.2 (11.8) | 77.5 (10.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 26.8 (2.0) | 28.5 (3.7) | 27.6 (3.0)
waist circumference [Mean (Standard Deviation); unit: cm] | 94.9 (4.5) | 99.8 (6.8) | 97.4 (6.2)
HbA1c [Mean (Standard Deviation); unit: percentage of HbA1c] | 6.1 (0.6) | 6.3 (1.8) | 6.2 (1.2)
fasting glucose [Mean (Standard Deviation); unit: mmol/l] | 5.5 (1.1) | 5.5 (2.2) | 5.5 (1.7)
HDL [Mean (Standard Deviation); unit: mmol/l] | 0.9 (0.2) | 0.8 (0.1) | 0.9 (0.2)
LDL [Mean (Standard Deviation); unit: mmol/l] | 2.8 (0.8) | 2.4 (0.9) | 2.6 (0.8)
insulin [Mean (Standard Deviation); unit: pmol/l] | 106.8 (65.8) | 84.5 (60.4) | 95.7 (62.5)
Triglyceride [Mean (Standard Deviation); unit: mmol/l] | 2.3 (1.1) | 1.5 (0.6) | 1.9 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Weight at 24 Weeks
Description: evaluate all participants' weight ，weight in kilograms
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: kilogram
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
kilogram | 0.2 (5.3) | -0.9 (3.1)

2. Secondary Outcome: Numbers of Participants Who Quit Smoking
Time Frame: 24 weeks
Measure: Number; unit: participants
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
participants | 0 | 0

3. Secondary Outcome: Changes From Baseline Craving for Nicotine Assessed by Visual Analog Scales (VAS) at 24 Weeks
Description: The visual analogue scale is a scale that is used to gauge smoking craving. Patients can choose a number from 0 to 10 to show their smoking craving, in which "0" represents "no craving" and "10" represents "intense urge".
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
score on a scale | -1.0 (2.9) | -1.9 (3.1)

4. Secondary Outcome: Depression Status Assessed by Self-rating Depression Scale（SDS）
Description: evaluate all participants' depression status by Self-rating depression scale（SDS)，which has a theoretical value range of 20-80. The SDS total score ranges, with the higher the score representing the higher level of severity of depression.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
score on a scale | 39.4 (8.2) | 33.6 (7.2)

5. Secondary Outcome: Anxiety Status Assessed by Self-Rating Anxiety Scale（SAS）
Description: evaluate all participants' depression status by Self-Rating Anxiety Scale，which has a theoretical value range of 20-80. The SAS total score ranges, with the higher the score representing the higher level of severity of anxiety.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
score on a scale | 31.1 (6.9) | 28.8 (4.2)

6. Secondary Outcome: Clinical Symptoms Assessed by the Positive and Negative Syndrome Scale (PANSS)
Description: Through a simple 40 to 50 minute talk with the patient, the physician scored 30 different symptoms on a scale of 1-7 to get their PANSS score. The total score range from 30-210. The PANSS total score ranges, with the higher the score representing the higher level of severity of clinical symptoms.
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
score on a scale | 52.5 (15.0) | 57.2 (18.9)

7. Secondary Outcome: Waist Circumference
Description: evaluate all participants' waist circumference，waist circumference in centimeters
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
cm | 98.6 (5.7) | 101.3 (6.6)

8. Secondary Outcome: Change in Fasting Blood Glucose Levels
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
mmol/l | 0.5 (1.5) | 1.0 (1.6)

9. Secondary Outcome: Change in Fasting Insulin Levels
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: pmol/l
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
pmol/l | 3.5 (74.4) | 11.0 (35.3)

10. Secondary Outcome: Change in Glycosylated Hemoglobin
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: percentage of hemoglobin
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
percentage of hemoglobin | 0.05 (0.6) | 0.4 (1.1)

11. Secondary Outcome: Change in Fasting Triglycerides Levels
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
mmol/l | -1.0 (0.9) | -0.4 (0.6)

12. Secondary Outcome: Change in Fasting HDL Cholesterol Levels
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
mmol/l | 0.0 (1.1) | 0.0 (0.1)

13. Secondary Outcome: Change in Fasting LDL Cholesterol
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: mmol/l
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
mmol/l | -0.4 (0.7) | -0.2 (0.7)

14. Secondary Outcome: Change in Leptin
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
ng/ml | 9.2 (5.9) | 10.6 (7.1)

15. Secondary Outcome: Change in Ghrelin
Time Frame: baseline and 24 weeks
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
Number analyzed (Participants) | 11 | 10
pg/ml | 352.2 (296.6) | 254.8 (106.4)

ADVERSE EVENTS:
Time Frame: The 24-week study time period
Arm/Group | Naltrexone and Bupropion | Placebo Naltrexone and Bupropion
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/10
Other Adverse Events (participants affected / at risk) | 6/11 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 4.76% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Naltrexone and Bupropion (N=11) | Placebo Naltrexone and Bupropion (N=10)
dry mouth (Gastrointestinal disorders) | 5 (5) | 0 (0)
mild abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
tachycardia (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-12-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT02736474/Prot_000.pdf
  • Statistical Analysis Plan (2015-12-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT02736474/SAP_001.pdf